CLINICAL TRIAL: NCT06839586
Title: The Efficacy and Safety of CMTS4520 for Chronic Diarrhoea in Adults： A Randomized, Double-Blind, Placebo-Controlled Trial.
Brief Title: CMTS4520 for Chronic Diarrhoea in Adults
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT-2024CMTS4520-003
Record Dates: First submitted 2025-02-14; First posted 2025-02-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-02

CONDITIONS: Diarrhoea
Keywords: CMTS4520; diarrhoea; randomized controlled trial; dietary fiber; probiotics
MeSH Terms: conditions — Diarrhea | interventions — Dietary Fiber; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The patient will receive CMTS4520 (dietary fiber probiotics) capsules daily for 4 weeks.
  Interventions: Drug: CMTS4520 (dietary fiber and probiotics)
- Control (Placebo Comparator): The patient will receive placebo of equal capsules daily for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CMTS4520 (dietary fiber and probiotics) — CMTS4520 is a synbiotic formulation containing a standardized ratio of plant-derived prebiotics and clinically validated probiotic strains. Participants will receive 4 weeks of CMTS4520 daily for chronic diarrhoea.
  Arms: Treatment
Drug: Placebo — Capsules with matching volume and consistent appearance to CMTS4520.
  Arms: Control

SUMMARY:
This is a randomized controlled trial to explore the efficacy and safety of CMTS4520 (Dietary Fiber Probiotics) for patients with chronic diarrhoea.

DETAILED DESCRIPTION:
At least 100 subjects who meet all the inclusion criteria but do not meet any exclusion criteria will be enrolled in this study. They will be randomly assigned to the CMTS4520 group (dietary fiber probiotics capsules) and the control group (placebo). Data of demographic characteristics, intestinal symptoms, medicine treatment usage and clinical outcomes will be collected. After treatment, they will enter the follow-up period for efficacy and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

Meet all of the following inclusion criteria :

1. Voluntary sign informed consent, age 18-70 years old (including the threshold), male and female.
2. Using the Rome IV criteria as the diagnostic criteria:

   1. Defecation frequency is greater than or equal to 3 times per day or significantly exceeds the usual habit, with a disease duration of > 4 weeks, or recurrent diarrhea with an intermittent period within 2 - 4 weeks;
   2. Loose stools: Types 5, 6, and 7 based on the Bristol Stool Form Scale.
3. The subject or his/her legal representative has given informed consent, is fully aware of the purpose of the study, is able to communicate well with the investigator, and is able to understand and comply with the requirements of the study.

Exclusion Criteria:

All exclusion criteria below are not met:

1. Participants with a history of intestinal resection.
2. Participants with organic lesions of the digestive tract (e.g., tumor, inflammation, anal fissures, Crohn's disease, ulcerative colitis, radiation enteritis, intestinal adhesions, intestinal tuberculosis) as confirmed by colonoscopy within the past 24 months.
3. Participants with diarrhoea secondary to systemic diseases affecting the digestive tract, including:

   1. Neurological diseases (e.g., Parkinson's disease, spinal cord injury, multiple sclerosis).
   2. Muscle diseases (e.g., amyloidosis, dermatomyositis).
   3. Psychiatric disorders or severe mood disorders (e.g., A Hospital Anxiety and Depression Scale score ≥15).
   4. Opioid-induced diarrhoea.
   5. Poorly controlled metabolic diseases (e.g., thyroid dysfunction) or metabolic diseases with gastrointestinal complications (e.g., gastrointestinal autonomic dysfunction, diabetic gastroparesis).
4. Diarrhea secondary to intestinal infectious diseases, including but not limited to Clostridioides difficile infection, chronic bacillary dysentery, intestinal tuberculosis, and parasitic infection-induced diarrhea.
5. Have a history of major surgery or severe trauma within 3 months and have not fully recovered.
6. Participants with any of the following cardiac abnormalities:

   1. New York Heart Association (NYHA) Class III or higher heart failure.
   2. Myocardial infarction or unstable angina within the past 6 months.
   3. Prolonged QTc interval on electrocardiogram (≥450ms for males, ≥470ms for females).
   4. Atrial arrhythmias that cannot be stably controlled by drugs and ventricular arrhythmias requiring pharmacological control (including grade 2 or higher atrioventricular block).
7. Participants with poor lung function, as assessed by the investigator, that may impact study treatment, such as acute chronic obstructive pulmonary disease(COPD) or those requring long-term oral, intravenous corticosteroids (excluding inhalant/spray formulations).
8. Uncontrolled immune diseases requring long-term systemic corticosteroid use (excluding topical use).
9. Participants with reproductive system disorders that may cause abdominal pain (e.g., ovarian cysts, endometriosis, primary dysmenorrhea).
10. Participants with significant laboratory abnormalities that, in the investigator's judgment, may affect safety or study completion, including:

    1. Hemoglobin <100g/L.
    2. Serum creatinine ≥1.5 times the upper limit of normal (ULN).
    3. Abnormal liver function (AST>1.5×ULN, ALT>1.5×ULN or total bilirubin >1.5×ULN).
    4. Clinically significant abnormalitieshe in routine stool tests or fecal occult blood indicating gastrointestinal lesions.
11. Participants with active hepatitis (requiring or undergoing long-term treatment), HIV, or active tuberculosis.
12. Participants with a history of drug or alcohol abuse (defined as consuming more than 14 standard drinks peer week: 1 standard drink= 360mL of beer, 45mL of 40% spirits, or 150mL of wine) or substance abuse.
13. Participants with known allergies or intolerances to the investigational drug, similar drugs or excipients.
14. Participants who have used anti-infective drugs (antibiotics, antifungals, antivirals) within 14 days prior to enrollment or require anti-infective treatment at the time of enrollment evaluation.
15. Participants who have used drugs or foods that regulate gut microbiota (e.g., bifidobacterium, probiotics, prebiotics, fermented milk, yogurt) within 2 weeks prior to screening or during the study.
16. Women who are pregnant, breastfeeding, or unwilling to use effective contraception for 3 months after the last dose of the study drug.
17. Participants who have participated in drug intervention clinical trials within 1 month prior to enrollment.
18. Any other condition that, in the investigator's judgment, makes the participant unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
The clinical response rate after treatment | One-week post-CMTS4520 administration，Two-week post-CMTS4520 administration，Four-week post-CMTS4520 administration，Eight-week post-CMTS4520 administration
  A clinical response was described as the change of the defecation frequency and the fecal consistency scores (assessed using the Bristol Stool Form Scale) after receiving CMTS4520.
  on the first day (D1) and the fourth week (D28) post-treatment compared to baseline, as well as the average weekly fecal consistency scores.

SECONDARY OUTCOMES:
The incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0 | Immediately post-CMTS4520 administration, One-week post-CMTS4520 administration，Two-week post-CMTS4520 administration，Four-week post-CMTS4520 administration，Eight-week post-CMTS4520 administration
  The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.).
The abdominal discomfort after treatment | One-week post-CMTS4520 administration，Two-week post-CMTS4520 administration，Four-week post-CMTS4520 administration，Eight-week post-CMTS4520 administration
  The scales include Gastrointestinal Symptom Rating Scale (GSRS) for abdominal discomfort.
The abdominal discomfort after treatment | One-week post-CMTS4520 administration，Two-week post-CMTS4520 administration，Four-week post-CMTS4520 administration，Eight-week post-CMTS4520 administration
  The scales include IBS Symptom Severity Scale (IBS-SSS) for abdominal discomfort.
The abdominal discomfort after treatment | One-week post-CMTS4520 administration，Two-week post-CMTS4520 administration，Four-week post-CMTS4520 administration，Eight-week post-CMTS4520 administration
  The scales include IBS Global Improvement Scale (IBS-GIS) for abdominal discomfort.
The quality of life after treatment | One-week post-CMTS4520 administration，Two-week post-CMTS4520 administration，Four-week post-CMTS4520 administration，Eight-week post-CMTS4520 administration
  IBS Quality of Life Scale (IBS-QOL) to measure quality of life.
The psychological states after treatment | One-week post-CMTS4520 administration，Two-week post-CMTS4520 administration，Four-week post-CMTS4520 administration，Eight-week post-CMTS4520 administration
  Hospital Anxiety and Depression Scale (HADS) to measure psychological states.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Department of Microbiota Medicine & Medical Centre for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Q, Verne ML, Fields JZ, Lefante JJ, Basra S, Salameh H, Verne GN. Randomised placebo-controlled trial of dietary glutamine supplements for postinfectious irritable bowel syndrome. Gut. 2019 Jun;68(6):996-1002. doi: 10.1136/gutjnl-2017-315136. Epub 2018 Aug 14. PMID 30108163
- [Background] Skrzydlo-Radomanska B, Prozorow-Krol B, Cichoz-Lach H, Majsiak E, Bierla JB, Kanarek E, Sowinska A, Cukrowska B. The Effectiveness and Safety of Multi-Strain Probiotic Preparation in Patients with Diarrhea-Predominant Irritable Bowel Syndrome: A Randomized Controlled Study. Nutrients. 2021 Feb 26;13(3):756. doi: 10.3390/nu13030756. PMID 33652763
- [Background] Weiss GA, Hennet T. Mechanisms and consequences of intestinal dysbiosis. Cell Mol Life Sci. 2017 Aug;74(16):2959-2977. doi: 10.1007/s00018-017-2509-x. Epub 2017 Mar 28. PMID 28352996
- [Background] Mari A, Abu Baker F, Mahamid M, Sbeit W, Khoury T. The Evolving Role of Gut Microbiota in the Management of Irritable Bowel Syndrome: An Overview of the Current Knowledge. J Clin Med. 2020 Mar 4;9(3):685. doi: 10.3390/jcm9030685. PMID 32143424
- [Background] Bhattarai Y, Muniz Pedrogo DA, Kashyap PC. Irritable bowel syndrome: a gut microbiota-related disorder? Am J Physiol Gastrointest Liver Physiol. 2017 Jan 1;312(1):G52-G62. doi: 10.1152/ajpgi.00338.2016. Epub 2016 Nov 23. PMID 27881403
- [Background] Lembo AJ, Lacy BE, Zuckerman MJ, Schey R, Dove LS, Andrae DA, Davenport JM, McIntyre G, Lopez R, Turner L, Covington PS. Eluxadoline for Irritable Bowel Syndrome with Diarrhea. N Engl J Med. 2016 Jan 21;374(3):242-53. doi: 10.1056/NEJMoa1505180. PMID 26789872
- [Background] Pimentel M, Lembo A, Chey WD, Zakko S, Ringel Y, Yu J, Mareya SM, Shaw AL, Bortey E, Forbes WP; TARGET Study Group. Rifaximin therapy for patients with irritable bowel syndrome without constipation. N Engl J Med. 2011 Jan 6;364(1):22-32. doi: 10.1056/NEJMoa1004409. PMID 21208106
- [Background] Peery AF, Dellon ES, Lund J, Crockett SD, McGowan CE, Bulsiewicz WJ, Gangarosa LM, Thiny MT, Stizenberg K, Morgan DR, Ringel Y, Kim HP, DiBonaventura MD, Carroll CF, Allen JK, Cook SF, Sandler RS, Kappelman MD, Shaheen NJ. Burden of gastrointestinal disease in the United States: 2012 update. Gastroenterology. 2012 Nov;143(5):1179-1187.e3. doi: 10.1053/j.gastro.2012.08.002. Epub 2012 Aug 8. PMID 22885331
- [Background] Camilleri M. Peripheral mechanisms in irritable bowel syndrome. N Engl J Med. 2013 Feb 7;368(6):578-9. doi: 10.1056/NEJMc1214185. No abstract available. PMID 23388017
- [Background] Enck P, Aziz Q, Barbara G, Farmer AD, Fukudo S, Mayer EA, Niesler B, Quigley EM, Rajilic-Stojanovic M, Schemann M, Schwille-Kiuntke J, Simren M, Zipfel S, Spiller RC. Irritable bowel syndrome. Nat Rev Dis Primers. 2016 Mar 24;2:16014. doi: 10.1038/nrdp.2016.14. PMID 27159638
- [Background] Farthing M, Salam MA, Lindberg G, Dite P, Khalif I, Salazar-Lindo E, Ramakrishna BS, Goh KL, Thomson A, Khan AG, Krabshuis J, LeMair A; WGO. Acute diarrhea in adults and children: a global perspective. J Clin Gastroenterol. 2013 Jan;47(1):12-20. doi: 10.1097/MCG.0b013e31826df662. No abstract available. PMID 23222211
- [Background] GBD 2021 Causes of Death Collaborators. Global burden of 288 causes of death and life expectancy decomposition in 204 countries and territories and 811 subnational locations, 1990-2021: a systematic analysis for the Global Burden of Disease Study 2021. Lancet. 2024 May 18;403(10440):2100-2132. doi: 10.1016/S0140-6736(24)00367-2. Epub 2024 Apr 3. PMID 38582094
- [Background] Sultana R, Luby SP, Gurley ES, Rimi NA, Swarna ST, Khan JAM, Nahar N, Ghosh PK, Howlader SR, Kabir H, Khan S, Jensen PKM. Cost of illness for severe and non-severe diarrhea borne by households in a low-income urban community of Bangladesh: A cross-sectional study. PLoS Negl Trop Dis. 2021 Jun 11;15(6):e0009439. doi: 10.1371/journal.pntd.0009439. eCollection 2021 Jun. PMID 34115764
- [Background] GBD 2016 Diarrhoeal Disease Collaborators. Estimates of the global, regional, and national morbidity, mortality, and aetiologies of diarrhoea in 195 countries: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Infect Dis. 2018 Nov;18(11):1211-1228. doi: 10.1016/S1473-3099(18)30362-1. Epub 2018 Sep 19. PMID 30243583
- [Background] GBD 2021 Diarrhoeal Diseases Collaborators. Global, regional, and national age-sex-specific burden of diarrhoeal diseases, their risk factors, and aetiologies, 1990-2021, for 204 countries and territories: a systematic analysis for the Global Burden of Disease Study 2021. Lancet Infect Dis. 2025 May;25(5):519-536. doi: 10.1016/S1473-3099(24)00691-1. Epub 2024 Dec 18. PMID 39708822
- [Background] Schiller LR, Pardi DS, Sellin JH. Chronic Diarrhea: Diagnosis and Management. Clin Gastroenterol Hepatol. 2017 Feb;15(2):182-193.e3. doi: 10.1016/j.cgh.2016.07.028. Epub 2016 Aug 2. PMID 27496381
- [Background] Arasaradnam RP, Brown S, Forbes A, Fox MR, Hungin P, Kelman L, Major G, O'Connor M, Sanders DS, Sinha R, Smith SC, Thomas P, Walters JRF. Guidelines for the investigation of chronic diarrhoea in adults: British Society of Gastroenterology, 3rd edition. Gut. 2018 Aug;67(8):1380-1399. doi: 10.1136/gutjnl-2017-315909. Epub 2018 Apr 13. PMID 29653941